CLINICAL TRIAL: NCT05500222
Title: A Randomized Double-blind Placebo-controlled Phase 3 Study to Evaluate the Effect of Resmetirom on Liver-related Outcomes in Patients With Well-compensated (Child-Pugh A) Non-alcoholic Steatohepatitis (NASH) Cirrhosis (MAESTRO-NASH-OUTCOMES)
Brief Title: A Phase 3 Study to Evaluate the Effect of Resmetirom on Clinical Outcomes in Patients With Well-compensated NASH Cirrhosis (MAESTRO-NASH-OUTCOMES)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Madrigal Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MGL-3196-19
Record Dates: First submitted 2022-08-11; First posted 2022-08-15 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: NASH; Cirrhosis, Liver
MeSH Terms: conditions — Liver Cirrhosis | interventions — resmetirom

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Resmetirom (Active Comparator): 80 mg daily
  Interventions: Drug: Resmetirom
- Placebo (Placebo Comparator): matching placebo daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Resmetirom — Randomized 80 mg
  Other Names: MGL-3196
  Arms: Resmetirom
Drug: Placebo — randomized matching placebo
  Arms: Placebo

SUMMARY:
This study will determine the effect of oral 80 mg resmetirom administered once daily on participants with well-compensated non-alcoholic steatohepatitis (NASH) cirrhosis by measuring the time to experiencing a Composite Clinical Outcome event.

DETAILED DESCRIPTION:
This is a multi-national, multicenter, double-blind, randomized, placebo-controlled study in participants with well-compensated NASH cirrhosis. Participants will be randomized 3:1 in a blinded manner to receive 80 mg resmetirom or matching placebo given orally once daily in the morning for the duration of the study (until the required number of Composite Clinical Outcome events are achieved). Composite Clinical Outcome events are defined as any of the following: liver-related and CV mortality, liver transplant, and significant hepatic events, including potential hepatic decompensation events (ascites, hepatic encephalopathy, or gastroesophageal variceal hemorrhage), and confirmed increase of Model for End-stage Liver Disease (MELD) score from <12 to ≥15. The study comprises an up to 60-day screening period and an approximately 3-year treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Definitive (by histologic documentation) or probable NASH as causative agent for cirrhosis, following a modified version of the NASH Cirrhosis: Liver Forum Consensus Definitions for Clinical Trials.
* a. Most recent biopsy (within last 5 years) shows cirrhosis with a NAS of ≥ 2, and at least two components: one being steatosis and at least one other component; OR NAS of ≥ 2, if steatosis = 0 or is ungraded with inflammation and/or ballooning, eligible with an MRI-PDFF >5%. If steatosis and ballooning and/or steatosis and inflammation are noted by the local pathologist, then the biopsy qualifies even if a NAS is not provided (Approximately 70% of the study patient population) b. Historical biopsy (within last 5 years) showed NASH with significant fibrosis with pathology report documenting "F2" or "F3", with at least steatosis either by biopsy with no minimal percentage required or by MRI-PDFF >5%, AND inflammation or ballooning. Now with cirrhosis, either by clinical history or current features, imaging, noninvasive tests, or biopsy (see Appendix 7) (Up to approximately 20% of study patient population) c. Historical biopsy (within last 5 years) shows steatosis. Pathology report documents steatosis with no minimal percentage required. Now with cirrhosis, either by clinical history or current features, imaging, noninvasive tests, or biopsy (see Appendix 7). Prescreening metabolic risk factors must include obesity and/or T2D. (Up to approximately 10% of study patient population.)
* Well-compensated NASH cirrhosis at screening and baseline with Child-Pugh A (score of 5-6) (no history of hepatic decompensation event).
* At least 3 metabolic risk factors
* Magnetic Resonance Imaging Proton Density Fat Fraction (MRI-PDFF) that is obtained during the Screening period or a historic MRI-PDFF at ≤8 weeks old at the time of randomization with no weight change ≥5% weight change in that interval.
* MRE ≥4.2 where MRE is available.
* Enhanced liver function (ELF) ≥9.8, only if MRE is unavailable or contraindicated.

Exclusion Criteria:

* Participants with a chronic liver diseases other than NASH cirrhosis, such as primary biliary cholangitis, primary sclerosing cholangitis, Hepatitis B positive, Hepatitis C, history or evidence of current active autoimmune hepatitis, history or evidence of Wilson's disease, history or evidence of alpha-1-antitrypsin deficiency, history or evidence of genetic hemochromatosis (hereditary, primary), evidence of drug-induced liver disease, as defined on the basis of typical exposure and history, known bile duct obstruction, or suspected or confirmed liver cancer, are excluded.
* Participants with MELD score ≥12 due to liver disease are excluded.
* Participants with a history of hepatic decompensation or impairment are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2022-08-26 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Incidence Of adjudicated Composite Clinical Outcome event | Baseline up to Month 36
  Any event of all-cause mortality, liver transplant, ascites, hepatic encephalopathy, gastroesophageal variceal hemorrhage, and confirmed increase of MELD score from <12 to >/= 15 due to liver disease

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Hare, Study Director — VP, Clinical Research
Locations (55):
- United States (53):
  - University of Alabama at Birmingham (UAB), Birmingham, Alabama
  - Arizona Liver Health - Chandler, Chandler, Arizona
  - Arizona Liver Health - Peoria, Peoria, Arizona
  - Adobe Clinical Research, Tucson, Arizona
  - Arizona Liver Health - Tucson, Tucson, Arizona
  - Arkansas Diagnostic Center/Liver Wellness Center, Little Rock, Arkansas
  - Arkansas Gastroenterology, North Little Rock, Arkansas
  - Southern California Research Center, Coronado, California
  - University of California, San Francisco-Fresno, Fresno, California
  - Univ. of California San Diego School of Medicine, La Jolla, California
  - Keck School of Medicine of USC, Los Angeles, California
  - California Liver Research Institute, Pasadena, California
  - South Denver Gastroenterology, Englewood, Colorado
  - Hi Tech and Global Research, Coral Gables, Florida
  - Top Medical Research Inc, Cutler Bay, Florida
  - Covenant Research - Fort Myers, Fort Myers, Florida
  - Nature Coast Clinical Research - Inverness, Inverness, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Ocala GI Research DBA Lake Center for Clinical Research, Lady Lake, Florida
  - Florida Research Institute, Lakewood Rch, Florida
  - Sanchez Clinical Research, Miami, Florida
  - Ocala GI Research, Ocala, Florida
  - St Johns Center for Clinical Research, Saint Augustine, Florida
  - Covenant Research, Sarasota, Florida
  - International Center for Research, Tampa, Florida
  - Florida Medical Clinic, Zephyrhills, Florida
  - Summit Clinical Research, Athens, Georgia
  - Gastrointestinal Specialists of Georgia, Marietta, Georgia
  - Kansas Medical Clinic - Gastroenterology, Topeka, Kansas
  - Delta Research Partners - Bastrop, Bastrop, Louisiana
  - Louisiana Research Center, Shreveport, Louisiana
  - Mercy Medical Center, Baltimore, Maryland
  - Kansas City Research Institute, Kansas City, Missouri
  - Premier Health Research, Sparta, New Jersey
  - Lucas Research, Morehead City, North Carolina
  - Regional Gastroenterology Associates of Lancaster, Flourtown, Pennsylvania
  - Rapid City Medical Center, Rapid City, South Dakota
  - Premier Medical Group, Clarksville, Tennessee
  - Gastro One, Cordova, Tennessee
  - Texas Clinical Research Institute, Arlington, Texas
  - Pinnacle Clinical Research - Austin, Austin, Texas
  - South Texas Research Institute - Brownsville, Brownsville, Texas
  - The Liver Institute at Methodist Dallas Medical Center, Dallas, Texas
  - Liver Center of Texas, Dallas, Texas
  - South Texas Research Institute - Edinburg, Edinburg, Texas
  - Pinnacle Clinical Research - Georgetown, Georgetown, Texas
  - Houston Research Institute, Houston, Texas
  - Pinnacle Clinical Research - San Antonio, San Antonio, Texas
  - Impact Research Institute, Waco, Texas
  - Digestive Health Research of Central Texas, Waco, Texas
  - GI Select Health Research, Richmond, Virginia
  - Hunter Holmes McGuire VA Medical Center, Richmond, Virginia
  - Liver Institute Northwest, Seattle, Washington
- Puerto Rico (2):
  - Latin Clinical Trials Center, San Juan
  - FDI Clinical Research (Fundacion de Investigacion de Diego), San Juan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Harrison SA, Ratziu V, Anstee QM, Noureddin M, Sanyal AJ, Schattenberg JM, Bedossa P, Bashir MR, Schneider D, Taub R, Bansal M, Kowdley KV, Younossi ZM, Loomba R. Design of the phase 3 MAESTRO clinical program to evaluate resmetirom for the treatment of nonalcoholic steatohepatitis. Aliment Pharmacol Ther. 2024 Jan;59(1):51-63. doi: 10.1111/apt.17734. Epub 2023 Oct 2. PMID 37786277